

| Official Title: | Impact of Behavioral Economic Strategies on Low-Income Older Adults' Food Choices in Online Retail Settings |
|---|---|
| NCT Number: | NCT04766034 |
| Study Number: | 20-01936 |
| Document Type: | Informed Consent Form |
| Date of the Document: | October 2, 2021 |

Study #: s20-01936 Version date: 9/23/2021 Page 1 of 1



## Research Subject Consent Form

You are being invited to take part in a research study about your diet and grocery shopping

behaviors. In Part 1, you will complete survey questions, which will take about 10 minutes.

In **Part 2**, you will also be asked to visit an online supermarket and select a typical week's worth of food for your household, which will take an **additional 10-15 minutes**. The shopping trip is only hypothetical, and no payment will be taken. You will be automatically entered into a lottery to have the items in your shopping cart delivered to your household for free. We will randomly select 100 participants to win this **extra incentive**.

To receive any incentives, you must complete the survey in Part 1 and the shopping trip task in Part 2.

Your participation in this study is voluntary and you can refuse to take part or stop at any time. There will be no costs to you for being in this study. Information collected and/or used for the purposes of this research will not be used by other researchers or distributed for future research studies.

There may be some minor risks from being in this study. You may experience frustration when answering questions. We take great care to protect your information but there is a slight risk of loss of privacy. You may not benefit personally from being in this study.

If you have any questions, you can email the Principal Investigator of this study Dr. Pasquale Rummo at pasquale.rummo@nyulangone.org or call 646-501-3371. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the NYU Grossman School of Medicine Institutional Review Board (IRB) at (212) 263-4110.

| Do you consent to take part in this research study and continue to the survey | ey? |
|---|---|
| □ Yes | |
| □ No | |